CLINICAL TRIAL: NCT00019708
Title: A Phase I and Pharmacologic Study of 17-(Allylamino)-17-Demethoxygeldanamycin (AAG, NSC 330507) in Adult Patients With Solid Tumors
Brief Title: Geldanamycin Analogue in Treating Patients With Advanced Solid Tumors or Non-Hodgkin's Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00819; NCI-2009-00819 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); UNMC 170-04; CDR0000066965; UNMC 170-04 (Other: University of Nebraska Medical Center); T98-0075 (Other: CTEP); NCT00001804 (obsolete NCT alias)
Record Dates: First submitted 2001-07-11; First posted 2003-01-27 (Estimated); Last update posted 2013-12-16 (Estimated); Status verified 2013-12

CONDITIONS: Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Nodal Marginal Zone B-cell Lymphoma; Non-Hodgkin Lymphoma; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Small Lymphocytic Lymphoma; Splenic Marginal Zone Lymphoma; Stage IV Adult Burkitt Lymphoma; Stage IV Adult Diffuse Large Cell Lymphoma; Stage IV Adult Diffuse Mixed Cell Lymphoma; Stage IV Adult Diffuse Small Cleaved Cell Lymphoma; Stage IV Adult Immunoblastic Large Cell Lymphoma; Stage IV Adult Lymphoblastic Lymphoma; Stage IV Grade 1 Follicular Lymphoma; Stage IV Grade 2 Follicular Lymphoma; Stage IV Grade 3 Follicular Lymphoma; Stage IV Mantle Cell Lymphoma; Stage IV Marginal Zone Lymphoma; Stage IV Small Lymphocytic Lymphoma; Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone; Lymphoma, Non-Hodgkin; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Mantle-Cell | interventions — tanespimycin

ARMS (1):
- Treatment (tanespimycin) (Experimental): Patients will receive infusions of tanespimycin analogue twice a week in weeks 1 and 3.
  Interventions: Drug: tanespimycin

INTERVENTIONS:
Drug: tanespimycin — Given IV
  Other Names: 17-AAG

SUMMARY:
Phase I trial to study the effectiveness of geldanamycin analogue in treating patients who have advanced solid tumors or non-Hodgkin's lymphoma. Drugs used in chemotherapy work in different ways to stop tumor cells from dividing so they stop growing or die.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose of geldanamycin analogue (AAG) in patients with advanced solid tumors.

II. To determine the toxic effects of this drug in this patient population. III. To determine the biochemical and molecular effects of this drug in normal and accessible tumor tissue in these patients.

IV. To determine the pharmacokinetics of this drug in these patients. V. To assess any antitumor activity of this drug in these patients.

OUTLINE: This is a dose-escalation study.

Patients receive geldanamycin analogue (AAG) IV over 1-6 hours once daily on days 1, 4, 15, and 18. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of AAG until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, an additional 10 patients are treated at the MTD.

Patients are followed every 6 weeks.

ELIGIBILITY:
Criteria:

* Platelet count at least 100,000/mm^3
* No leukemia
* No active CNS involvement with tumor
* ECOG 0-2
* Life expectancy: at least 3 months
* Absolute neutrophil count at least 2,000/mm^3
* No New York Heart Association class III or IV heart failure
* No history of myocardial infarction within the past year
* Bilirubin =< upper limit of normal (ULN)
* AST no greater than 2 times ULN (no greater than 98 U/L)
* No uncontrolled dysrhythmias
* No poorly controlled angina
* No serious ventricular arrhythmia (i.e., ventricular tachycardia (VT) or ventricular fibrillation (VF) >= 3 beats in a row)
* QTc interval =< 450 msec for men or =< 470 msec for women
* LVEF >= 40% by MUGA
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* No other serious medical condition that would preclude study participation
* No serious hypersensitivity to egg products
* No concurrent anticancer immunotherapy
* At least 4 weeks since prior chemotherapy and recovered
* No other concurrent anticancer chemotherapy (e.g., cyclophosphamide, doxorubicin, vincristine, and prednisone [CHOP] or mechlorethamine, vincristine, procarbazine, and prednisone [MOPP])
* No concurrent anticancer hormonal therapy
* Concurrent glucocorticoids as antiemetics for nonmalignant disease allowed
* At least 4 weeks since prior radiotherapy and recovered
* No concurrent radiotherapy
* No concurrent major surgery
* No concurrent anticancer glucocorticoids
* Creatinine =< ULN or Creatinine clearance at least 60 mL/min
* No concurrent medications that cause QTc prolongation
* Histologically confirmed advanced solid tumor for which no curative therapy exists
* Non-Hodgkin's lymphoma allowed
* No concurrent drugs that interfere with hepatic CYP3A4 metabolism (e.g., grapefruit juice, ketoconazole, fluconazole, itraconazole, cyclosporine, erythromycin, clarithromycin, cimetidine, terfenadine, astemizole, indinavir, or nelfinavir mesylate)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 1999-06; Primary Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of tanespimycin | 28 days
  DLT are defined as any greater than or equal to grade 3 non-hematologic toxicity (except for alopecia of any grade, grade 3 nausea or vomiting during less than maximal antiemetic therapy, and grade 3 fever in the absence of neutropenia and infection), any grade 4 hematologic toxicity (except for anemia of any grade), or the inability to resume treatment by day 42 (longer than two week delay) because of drug related toxicity.

SECONDARY OUTCOMES:
Biomolecular effects of tanespimycin in normal tissues such as peripheral blood and bone marrow mononuclear cells | Up to day 5
  Changes in the protein expression of the molecular markers will be assessed by western blot analysis.
Pharmacokinetics of tanespimycin | Pre-infusion, 20 minutes, 40, 50, 60 (end of infusion), 70, 80, 95 and 110 minutes, and 2.5, 3, 4, 5, 6.5, 8, 10, 14 and 24 hours
  Determined by HPLC with photodiode array detection. The pharmacokinetic parameters that will be determined for parent drug include the maximum plasma concentration (Cmax), time of maximum plasma concentration (Tmax), area under the concentration-time curve (AUC), terminal half-life, clearance and volume of distribution.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Grem, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States